CLINICAL TRIAL: NCT03236688
Title: Detection of ARv7 in the Plasma of Men With Advanced Metastatic Castrate Resistant Prostate Cancer (MCRP)
Status: Suspended | Type: Observational
Sponsor: Exosome Diagnostics, Inc. (Industry)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: ECT2015-004
Record Dates: First submitted 2016-02-23; First posted 2017-08-02 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Metastatic Castrate Resistant Prostate Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 10-20 mL of whole blood collected in K2EDTA Plasma Preparation Tubes (PPT) will be acquired via standard venipuncture and processed to plasma.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MCRPC: Metastatic Castrate Resistant Prostate Cancer (MCRPC) Patients

SUMMARY:
Demonstrate detection of ARv7 splice variant transcripts from exosomes in the circulation of MCRPC patients pre and post treatment with selective Androgen pathway inhibitors (i.e. abiraterone and enzalutamide)

DETAILED DESCRIPTION:
Primary Objective

-Demonstrate detection of ARv7 splice variant transcripts from exosomes in the circulation of MCRPC patients pre and post treatment with selective Androgen pathway inhibitors (i.e. abiraterone and enzalutamide)

Secondary and Exploratory Objectives

* Correlate ARv7 status with PSA response (>/=50% decline in PSA level from baseline, maintained for >/=4 weeks) at any time after the initiation of therapy.
* Comparison of median progression free survival (PFS) and overall survival (OS).
* Determine additional molecular lesions in exoRNA and cfDNA in MCRPC patients post-treatment with androgen pathway inhibitors.
* Correlate other AR-variants (non ARv7) with clinical outcomes including PSA response.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have histologically confirmed diagnosis of adenocarcinoma of the prostate.
2. Clinical or radiographic evidence of metastatic disease.
3. Planned therapy with either enzalutamide or abiraterone acetate within the coming 6 weeks.
4. Evidence of disease progression on or following most recent therapy as evidenced by the following:

   * Radiographic evidence of disease progression as defined by one or more new bone scan lesions.
   * Growth of soft tissue / visceral metastases to greater than one centimeter in longest diameter.
   * Progressive disease despite 'castration levels' of serum testosterone (<50ng/dL with continued androgen deprivation therapy.
5. At least two of the following high risk features during screening for rapid disease progression:

   * Anemia with a hemoglobin <12.0 g/dL
   * Elevated alkaline phosphatase
   * High lactate dehydrogenase (LDH)
   * Presence of visceral metastasis on imaging
   * Presence of clinically significant pain requiring opioid analgesics.
   * PSA doubling time under 3 months on most recent therapy
   * PSA values obtained 2 or more weeks apart, with last value being 2.0ng/mL or higher.
6. Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

1. Receiving or intend to receive concurrent chemotherapy
2. Hepatitis (all types) in patient's medical record
3. HIV documented in patient's medical record
4. History of intercurrent or past medical history or psychiatric illness that would make participation in a blood drawing protocol difficult or not feasible.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-02; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Detection of ARv7 splice variant in the circulation of MCRPC patients. PSA response rate in ARv7 positive patients. | Two years
  The detection of ARv7 splice variants in samples will be considered both binary: positive or negative/not assessable and level based. ARv7 splice variants from exosomes will be detectable from baseline in 50% of both API; PSA response rates will be 10% or less in ARv7 positive patients. With a sample of 30 patients (as reported in the NEJM study) per cohort would allow the study to have an 85% power to detect a difference of 50 percentage points in PSA response rates, with the use of a two-sided test at an alpha level of 0.1.

SECONDARY OUTCOMES:
Detection of ARv7 splice variant in the circulation of MCRPC patients. PSA response rate in ARv7 negative patients. | Two years
  The detection of ARv7 splice variants in samples will be considered both binary: positive or negative/not assessable and level based. ARv7 splice variants from exosomes will be detectable from baseline in 50% of both API; PSA response rates will be 50% or more in ARv7 negative patients. With a sample of 30 patients (as reported in the NEJM study) per cohort would allow the study to have an 85% power to detect a difference of 50 percentage points in PSA response rates, with the use of a two-sided test at an alpha level of 0.1.

CONTACTS AND LOCATIONS:
Overall Officials: Roger Tun, Study Director — Exosome Diagnostics, Inc.
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided